CLINICAL TRIAL: NCT01779947
Title: An Investigator-Blind, Randomized, Parallel-Group, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Bioequivalence of Estradiol Vaginal Inserts, USP 10 mcg and Vagifem® (Estradiol Vaginal Tablets) 10 mcg and Compare Both Active Treatments to a Placebo Control in Female Subjects With Moderate to Severe Symptoms of Vulvar and Vaginal Atrophy Associated With Menopause
Brief Title: Study to Evaluate the Safety and Bioequivalence of Estradiol Vaginal Inserts, 10 mcg and Vagifem® 10 mcg and Compare to Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amneal Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AM-ESD-001
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Atrophic Vaginitis Due to Menopause
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Estradiol Vaginal Insert 10 mcg (Experimental): Estradiol Vaginal Insert 10 mcg - Test Product
  Interventions: Drug: Estradiol Vaginal Tablets 10 mcg
- Vagifem Tablets 10 mcg (Active Comparator): Vagifem® (Estradiol Vaginal Tablets) 10 mcg - Reference Listed Drug
  Interventions: Drug: Estradiol Vaginal Tablets 10 mcg
- Placebo (Placebo Comparator): Placebo for the test product Estradiol Vaginal Tablets 10 mcg
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Estradiol Vaginal Tablets 10 mcg
  Other Names: Vagifem®
  Arms: Estradiol Vaginal Insert 10 mcg; Vagifem Tablets 10 mcg
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety and efficacy of generic Estradiol Vaginal Inserts, USP 10 mcg to the reference product Vagifem® 10 mcg and to determined whether the efficacy of each of the 2 active treatments is superior to that of the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide and understand written informed consent for the study.
* Healthy female subject aged 30 to 75 years, inclusive, who was postmenopausal, defined as having had 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) levels > 40 mIU/mL, or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* At least 1 subject-assessed moderate to severe symptom of VVA among the following 4 symptoms that was identified by the subject as being most bothersome to her:
* Vaginal dryness
* Vaginal and/or vulvar irritation/itching
* Dysuria
* Vaginal pain associated with sexual activity OR
* The presence of vaginal bleeding associated with sexual activity
* Had ≤ 5% superficial cells on vaginal smear cytology at Visit 1.
* Vaginal pH > 5.0 at Visit 1.
* Systolic blood pressure ≤ 150 mm Hg and diastolic blood pressure ≤ 90 mm Hg at Visit 1.
* If > 40 years old, documentation of a negative mammogram (obtained at Visit 1 or within 9 months prior to Visit 1). A radiology report documenting a negative mammogram must have been available and must have been taken within 9 months of Visit 1 or obtained at Visit 1.
* Normal clinical breast examination at Visit 1.
* For women with intact uterus, vaginal ultrasonography confirmation at Visit 1 of an inactive endometrial lining, with an endometrial thickness < 4 mm.
* Documented Pap smear conducted within the previous 12 months of Visit 1 with no findings that the investigator believed would contraindicate the use of topical vaginal estradiol.
* In general good health with no clinically significant disease other than symptoms of VVA that might have interfered with the study evaluations.
* Was willing and able to understand and comply with the requirements of the study, including applying the medication as instructed, returning for the required study visits, complying with therapy prohibitions, and able to complete the study.

Exclusion Criteria:

* Known hypersensitivity to estradiol vaginal tablet or any component of the study medication.
* A subject who had received any treatment listed below more recently than the indicated washout period prior to Visit 1/Screening/Baseline.
* Prohibited Medications - (Washout Period Prior to Visit 1/Screening/Baseline)
* Vaginal lubricants or moisturizers - (at least 48 hours (2 days))
* Vaginal hormonal products (rings, creams, gels) - (at least 1 week (7 days))
* Transdermal estrogen alone or estrogen/progestin products - (at least 4 weeks (28 days))
* Oral estrogen and/or progestin therapy - (at least 8 weeks (56 days))
* Intrauterine progestin therapy - (at least 8 weeks (56 days))
* Progestin implants and estrogen alone injectable drug therapy - (at least 3 months (90 days))
* Estrogen pellet therapy or progestin injectable drug therapy - (at least 6 months (180 days))
* Subject who had engaged in sexual intercourse within 48 hours (2 days) of Visit 1.
* Screening mammogram or clinical breast examination results indicating any suspicion of breast malignancy.
* History of undiagnosed vaginal bleeding.
* Known bleeding disorder.
* History of significant risk factors for endometrial cancer (i.e., tamoxifen use, prior pelvic radiation therapy, and endometrial hyperplasia).
* For women with an intact uterus, screening vaginal ultrasonography showing endometrial thickness of ≥ 4 mm.
* Known, suspected, or history of breast cancer or cervical cancer.
* Known or suspected estrogen-dependent neoplasia.
* History of uncontrolled hypertension.
* Active deep vein thrombosis, pulmonary embolism, or history of these conditions.
* Active arterial thromboembolic disease (e.g., stroke or myocardial infarction) or a history of these conditions.
* Known liver dysfunction or disease.
* Known anaphylactic reaction or angioedema to estradiol vaginal tablets.
* Known protein C, protein S, antithrombin deficient, or other known thrombophilic disorders. - Active vaginal herpes simplex infection or any known concurrent vaginal infections.
* Abnormal Pap smear within the previous 12 months of Visit 1 or obtained during Visit 1. Any evidence of malignancy or premalignant changes or atypical squamous cell of undetermined significance (ASCUS) Pap smear with positive high risk human papillomavirus (HPV).
* Any clinically significant condition or situation (including laboratory values) other than the condition being studied that, in the opinion of the investigator, would have interfered with the study evaluations or optimal participation in the study.
* Use of any investigational drugs or device within 30 days of signing the ICF.
* Current participation in any other clinical study involving an investigational drug or device.
* Consumed excessive amounts of alcohol, abused drugs, or had any condition that would have compromised compliance with this protocol.
* Previous participation in this study.
* Subjects who, in the opinion of the Investigator, would have been non-compliant with the requirements of the study protocol.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Responders | Day 15 (1 day after the administration of the 14th dose of study treatment)
  A responder was defined as a subject with at least a 25% reduction from baseline in the sum of % basal/parabasal and % intermediate cells on vaginal cytology AND vaginal pH < 5.0 with a change from baseline vaginal pH of at least 0.5, where baseline values were collected at Visit 1

SECONDARY OUTCOMES:
Treatment Success | Day 15
  Treatment success was defined as a subject who achieved a score of 0 (none) or 1 (mild) at Visit 3 for the Most Bothersome Symptom (MBS) if her MBS was vaginal dryness, vaginal or vulvar irritation or itching, dysuria or vaginal pain associated with sexual activity, or a result of absence (0) at Visit 3 if her MBS was vaginal bleeding with sexual activity.

CONTACTS AND LOCATIONS:
Overall Officials: W. Todd Kays, PhD, Study Chair — Amneal Pharmaceuticals, LLC
Locations (25):
- United States (25):
  - Medical Affiliated Research center, Inc., Huntsville, Alabama
  - Montogmery Women's Health Associates, Montgomery, Alabama
  - Medical Center for Clinical Research, San Diego, California
  - Women's Health Care Research Corp., San Diego, California
  - Downtown Women's Health care, Denver, Colorado
  - Horizons Clinical Research Center, Denver, Colorado
  - James A. Simon, MD PC/ Women's Health and Research Consultants, Washington D.C., District of Columbia
  - Visions Clinical Reserach, Boynton Beach, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Altus Research, Lake Worth, Florida
  - New Age Medical Reserach Group, Miami, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Atlanta North Gynecology, Roswell, Georgia
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Cypress Medical Research Center. LLC, Wichita, Kansas
  - Meridian Health Care, Neptune City, New Jersey
  - Center for Women's Health and Wellness, LLC/ Women's Health Research Center, Plainsboro, New Jersey
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Lyndhurst Clinical Research, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Hawthorne Medical Research, Inc., Winstom-Salem, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Columbus Center for Women;s Health Reserach, Columbus, Ohio
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Seatlle Womne's Health,Reserach, Gynecology, Seattle, Washington